CLINICAL TRIAL: NCT03138031
Title: Outcome of Percutaneous Ethanol Alcohol Injection (PEI) for the Large and Unresectable Hepatocellular Carcinoma.
Brief Title: Percutaneous Ethanol Alcohol Injection for the Large and Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Ribat University (Other)
Responsible Party: Principal Investigator, Osama Mohamed Elsanousi, General Surgeon, The National Ribat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS-002-17
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Percutaneuos Ethanol alcohol injection
MeSH Terms: interventions — Ethanol; Injections

STUDY DESIGN:
Intervention Model Description: Single Group Assignment. Prospective and non-randomized clinical trial
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous Ethanol Injection (PEI) (Experimental): Those participants receive percutaneous ethanol alcohol injection for the large and unresectable HCC. Absolute alcohol; weekly sessions; under close monitoring; maximum of 30 mls; no anaesthesia needed and a maximum pain score of "8" during the procedure. Postprocedure analgesia may be required.
  Interventions: Procedure: Percutaneous ethanol alcohol injection

INTERVENTIONS:
Procedure: Percutaneous ethanol alcohol injection — Day-case procedure; weekly sessions; uses absolute alcohol; under close monitoring; maximum dose of 30 ml; no anesthesia needed and a maximum pain score of "8" limits the procedure. Post-procedure analgesia may be required.

SUMMARY:
Assessment of the long-term outcome of percutaneous ethanol alcohol injection (PEI) for the large and unresectable hepatocellular carcinoma: single center non-randomized trial.

DETAILED DESCRIPTION:
Assessment of the overall (OS); one year; two years and three years' survival rates; the disease free survival (DFS) and the tumor response rate in the patients undergoing (PAT or PEI) for the large and inoperable hepatocellular carcinoma. This is a prospective non randomized trial carried out at the Ribat University Hospital between May 2017 to April 2020.

ELIGIBILITY:
Inclusion Criteria:

* Review and sign informed consent;
* Between 15 and 80 years of age at time of trial enrollment;
* Documented pathological and/or radiological diagnosis of hepatocellular carcinoma;
* Radiologically documented tumor size of > 5 centimeters;
* Radiologically documented liver cirrhosis.

Exclusion Criteria:

* American Anesthesia Association (ASA) Class IV or V and/or any
* contraindications to general anesthesia;
* Uncontrollable ascites;
* Deep persistent jaundice;
* Hepatic encephalopathy;
* Coagulopathy;
* Severe thrombocytopenia;
* Unable or unwilling to attend follow up visits and examinations;
* Other associated surgical procedure;

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 3 years
  The percentage of HCC patients who are still alive for three years after they started PEI for HCC.

SECONDARY OUTCOMES:
Disease free survival | 3 years
  Percentage of HCC patients who are alive and well (without a recurrence of their HCC) 3 years after PEI.
Major complications' rate | 3 years
  Incidence of post-procedure Common Terminology Criteria for Adverse Events (CTCAE v4.03) grade
Tumor response rate | 3 years
  Mean percentage reduction in the sizes of the patients' tumors

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Elsanousi, MD, Principal Investigator — The National Ribat University; Murtada M Mohamed, MD, Principal Investigator — Ribat University Hospital
Locations (1):
- Ribat University Hospital, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: No